CLINICAL TRIAL: NCT03874182
Title: Prevalence of Dental Traumatic Injuries in A Group of Egyptian Children With Special Health Care Needs Aging 6-14 Years : A Cross -Sectional Study
Brief Title: Prevalence of Dental Traumatic Injuries in A Group of Egyptian Children With Special Health Care Needs
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sara Refaat Ahmad, Principle investigator, Cairo University
Other Study IDs: 1.2
Record Dates: First submitted 2019-03-12; First posted 2019-03-14 (Actual); Last update posted 2019-04-22 (Actual); Status verified 2019-03

CONDITIONS: Dental Trauma
Keywords: Prevalence; Dental trauma; Special health care needs children

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A cross-sectional descriptive study which will investigate the Prevalence of Dental Traumatic injuries in A Group of Egyptian Children with Special Health Care needs aging 6-14 years Attending Pediatric Dentistry and Dental Public Health Department at Faculty of Dentistry, Cairo University., Investigate the types, causes, and possible risk factors and treatment sought.

DETAILED DESCRIPTION:
Study Design:A Cross -sectional descriptive study design. Participant: Children with special health care needs between 6 to 14 years. Setting: Patients coming to pediatric dentistry and dental public health department in Cairo University.

All the procedures will be explained to the parents or guardians prior to the investigation.An informed consent will be signed by parents.

Method:Data for the study will be collected using an interviewer - administered questionnaire.The interviewer - administered questionnaire will be in Arabic in multiple choice form and will include:

1. History of current and previous dental trauma: including place and cause of the trauma.
2. Treatment sought :

If treatment was sought, the parent will be asked to indicate the type of treatment received:

1. Pharmacological: prescription of pain killers, antibiotics, and tetanus injections.
2. Dental: restorative, endodontic, surgical, prosthetic, and splinting.

If treatment was not sought, the parent will be asked to select one or more of the reasons for this, including the following:

1. Financial: transportation, dental insurance coverage, and acceptance of insurance by dentist.
2. Parental attitude: lack of trust in dentists, inability to wait for appointment, lack of dental awareness such as not knowing where to go, or the belief that the trauma was not worth seeking treatment.
3. Difficulties in getting an appointment: availability of dental clinics that was willing to see the children.

The clinical examination will be carried out under artificial light of dental unit by using mirror and Goldman- Fox periodontal probe according to custom-made examination chart which is made according to Assessment of acute traumatic injuries chart (Adopted from American Academy of Pediatric Dentistry, Pediatr Dent 24 (7suppl):95-96, 2002) and consisted of:

* Child's demographic data (Personal history), past and present medical history, past dental history and history of the trauma.
* Extra oral examination and intra oral examination to detect:

  1. The presence/absence of dental traumatic injuries determined by direct clinical examination, when trauma is present will be recorded according to the Andreasen classification (1994) .
  2. Condition of the injured tooth: mobility, tenderness to percussion, and discoloration of traumatized teeth.
  3. Possible associated risk factors with dental traumatic injuries: overjet, overbite, lip competence, anterior crowding.
  4. Using Goldman -Fox periodontal probe overjet will be measured as the amount of extension of the incisal edges of upper incisors labially beyond the incisal edges of the lower incisors when the jaws are closed normally. Overbite will be measured as the amount of overlap of the incisal edges of the upper anterior teeth and the incisal edges of the lower teeth when the jaws are closed.
* Dental photographs

ELIGIBILITY:
Inclusion Criteria:

* Age of children between 6 and 14 years old
* Both sexes.
* Patient who has one of the following conditions:

  * Cerebral palsy
  * Down's syndrome
  * Neurobehavioral disorders such as autism spectrum disorder (ASD) and attention deficient hyperactive disorder( ADHD)
  * Intellectual disability and learning difficulties
  * Motor difficulty
  * Visual impairment
  * Hearing and speech impairment
  * Multiple disability : patients with more than one medical condition
  * Developmental Delay and Epilepsy

Exclusion Criteria:

* Parent refusal to join the study
* Patient with non specified condition

Ages: 6 Years to 14 Years | Sex: All
Age Groups: Child
Study Population: This cross-sectional study included a convenient sample from all patients with special health care needs coming to pediatric dentistry and dental public health department in Cairo University.
Sampling Method: Non-Probability Sample
Enrollment: 763 (Estimated)
Dates: Start 2019-05 (Estimated); Primary Completion 2020-05 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Prevalence of dental traumatic injuries in children with special health care needs | Data collection will be performed within one year from the starting date of the study
  Through clinical examination to detect presence or absence of dental trauma will detect presence/absence of dental trauma

SECONDARY OUTCOMES:
Types of dental traumatic injuries | Data collection will be performed within one year from the starting date of the study
  Through clinical examination when trauma is present will be recorded according to the Anderson's classification (1994) Clinical examination
Causes of dental traumatic injuries | Data collection will be performed within one year from the starting date of the study
  History of the causes of dental trauma will be obtained through an interviewer - administered questionnaire which will be in Arabic and the questions in multiple choice form
Risk factors of dental traumatic injuries | Data collection will be performed within one year from the starting date of the study
  Overjet, overbite, lip competence, anterior crowding. Using Goldman -Fox periodontal probe overjet will be measured as the amount of extension of the incisal edges of upper incisors labially beyond the incisal edges of the lower incisors when the jaws are closed normally. Overbite will be measured as the amount of overlap of the incisal edges of the upper anterior teeth and the incisal edges of the lower teeth when the jaws are closed

IPD SHARING:
Plan to Share IPD: Undecided